CLINICAL TRIAL: NCT02306421
Title: A Multi Center Clinical Trial of the Efficacy and Safety of Rph With the Simplified Milligan-Morgan Surgery on Treatment of Mixed Hemorrhoids
Brief Title: A Multi Center Clinical Trial of Rph With the Simplified Milligan-Morgan Surgery on Treatment of Mixed Hemorrhoids
Acronym: RPHSMMH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Second Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other)
Collaborators: Hunan University of Traditional Chinese Medicine (Other); Zhengfeng Medical Technology Company Limited of Hunan Province (Industry)
Responsible Party: Principal Investigator, YONG-HENG HE, Study Director、Professor, The Second Affiliated Hospital of Hunan University of Traditional Chinese Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SecondUTCM
Record Dates: First submitted 2014-08-24; First posted 2014-12-03 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-11

CONDITIONS: Mixed Hemorrhoids
Keywords: RPH with the simplified Milligan-Morgan surgery; mixed hemorrhoids; the effectiveness and safety; A multi center clinical trial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- RPH with the simplified Milligan-Morgan (Active Comparator): RPH is a new therapy for hemorrhoid following the improvement of rubber band ligation. The treatment principle is: shrinkage of mucous membrane after the ligation, lift of anal cushion, the local inflammatory response resulting in adhesion of mucosa and submucosa and shallow muscle layer, anal cushion fixing to a higher position, at the same time by using the elastic contraction of automatic elastic line partly blocking blood supply of Internal hemorrhoids or reducing venous stasis, decreasing congestion hypertrophy of hemorrhoids. Simplified Milligan-Morgan is a surgical option which was improved and developed by Professor He,well-known traditional Chinese doctor from Hunan province, based on Milligan-Morgan in 1971.The operation method is simple, the operation time is shortened.
  Interventions: Procedure: RPH with the simplified Milligan-Morgan
- PPH with the simplified Milligan-Morgan (Active Comparator): According to anal cushion down theory of the formation of hemorrhoids, the Italy scholar Longo pioneered a new method for the treatment of circular prolapsed internal hemorrhoids In 1998.Its principle is resection of lower rectal mucosa and submucosa of the intestinal wall tissue in the ring above the hemorrhoids through surgical staples,anastomosis of the proximal and distal mucosa , lifting and fixing down anal cushion, recovering to the normal anatomical position.Simplified Milligan-Morgan is a surgical option which was improved and developed by Professor He,well-known traditional Chinese doctor from Hunan province, based on Milligan-Morgan in 1971.The operation method is simple, the operation time is shortened.
  Interventions: Procedure: PPH with the simplified Milligan-Morgan
- R P H (Active Comparator): RPH is a new therapy for hemorrhoid following the improvement of rubber band ligation.The treatment principle is: shrinkage of mucous membrane after the ligation, lift of anal cushion, the local inflammatory response resulting in adhesion of mucosa and submucosa and shallow muscle layer , anal cushion fixing to a higher position, at the same time by using the elastic contraction of automatic elastic line partly blocking blood supply of Internal hemorrhoids or reducing venous stasis, decreasing congestion hypertrophy of hemorrhoids , making hemorrhoidal lump shrink, thus eliminating bleeding and prolapse symptoms of hemorrhoid.It is suitable for internal hemorrhoids in every period and internal hemorrhoids part of mixed hemorrhoid.
  Interventions: Procedure: RPH
- P P H (Active Comparator): According to anal cushion down theory of the formation of hemorrhoids, the Italy scholar Longo pioneered a new method for the treatment of circular prolapsed internal hemorrhoids-PPH.In 1998.Its principle is resection of lower rectal mucosa and submucosa of the intestinal wall tissue in the ring above the hemorrhoids through surgical staples,anastomosis of the proximal and distal mucosa , lifting and fixing down anal cushion, recovering to the normal anatomical position
  Interventions: Procedure: PPH
- Milligan-Morgan (Active Comparator): Milligan-Morgan surgery ,created in 1937 by Milligan etc,whose essence is to excise hemorrhoids of increasing prolapse in anatomy has good curative effect, low recurrence.It is currently the most common clinical surgery.
  Interventions: Procedure: Milligan-Morgan

INTERVENTIONS:
Procedure: RPH with the simplified Milligan-Morgan — RPH is a new therapy for hemorrhoid following the improvement of rubber band ligation. The treatment principle is: shrinkage of mucous membrane after the ligation, lift of anal cushion, the local inflammatory response resulting in adhesion of mucosa and submucosa and shallow muscle layer, anal cushion fixing to a higher position, at the same time by using the elastic contraction of automatic elastic line partly blocking blood supply of Internal hemorrhoids or reducing venous stasis, decreasing congestion hypertrophy of hemorrhoids. Simplified Milligan-Morgan is a surgical option which was improved and developed by Professor He,well-known traditional Chinese doctor from Hunan province, based on Milligan-Morgan in 1971.The operation method is simple, the operation time is shortened.
  Arms: RPH with the simplified Milligan-Morgan
Procedure: PPH with the simplified Milligan-Morgan — According to anal cushion down theory of the formation of hemorrhoids, the Italy scholar Longo pioneered a new method for the treatment of circular prolapsed internal hemorrhoids In 1998.Its principle is resection of lower rectal mucosa and submucosa of the intestinal wall tissue in the ring above the hemorrhoids through surgical staples,anastomosis of the proximal and distal mucosa , lifting and fixing down anal cushion, recovering to the normal anatomical position.Simplified Milligan-Morgan is a surgical option which was improved and developed by Professor He,well-known traditional Chinese doctor from Hunan province, based on Milligan-Morgan in 1971.The operation method is simple, the operation time is shortened.
  Arms: PPH with the simplified Milligan-Morgan
Procedure: RPH — RPH is a new therapy for hemorrhoid following the improvement of rubber band ligation.The treatment principle is: shrinkage of mucous membrane after the ligation, lift of anal cushion, the local inflammatory response resulting in adhesion of mucosa and submucosa and shallow muscle layer , anal cushion fixing to a higher position, at the same time by using the elastic contraction of automatic elastic line partly blocking blood supply of Internal hemorrhoids or reducing venous stasis, decreasing congestion hypertrophy of hemorrhoids , making hemorrhoidal lump shrink, thus eliminating bleeding and prolapse symptoms of hemorrhoid.It is suitable for internal hemorrhoids in every period and internal hemorrhoids part of mixed hemorrhoid.
  Arms: R P H
Procedure: PPH — According to anal cushion down theory of the formation of hemorrhoids, the Italy scholar Longo pioneered a new method for the treatment of circular prolapsed internal hemorrhoids In 1998.Its principle is resection of lower rectal mucosa and submucosa of the intestinal wall tissue in the ring above the hemorrhoids through surgical staples,anastomosis of the proximal and distal mucosa , lifting and fixing down anal cushion, recovering to the normal anatomical position
  Arms: P P H
Procedure: Milligan-Morgan — Milligan-Morgan surgery ,created in 1937 by Milligan etc,whose essence is to excise hemorrhoids of increasing prolapse in anatomy has good curative effect, low recurrence.It is currently the most common clinical surgery.
  Arms: Milligan-Morgan

SUMMARY:
Simplified Milligan-Morgan is a surgical option which was improved and developed by Professor He,well-known traditional Chinese doctor from Hunan province,based on Milligan-Morgan.RPH is a new therapy for hemorrhoid following the improvement of rubber band ligation.RPH +Simplified Milligan-Morgan is one of important means of modern surgery.The operation method was improved and developed on the basis of Chinese medicine traditional loop ligature and it also embodies uniqueness and advantage of the treatment of mixed hemorrhoids combined traditional Chinese and Western Medicine.The study intends to compare five surgery ways through 3000 cases of patients with mixed hemorrhoid from 12 hospitals,observing the efficacy and safety of various operative methods.Exploration of RPH + Simplified Milligan-Morgan operation indication, contraindication, operation steps and key points, and the operation complications and sequelae and treatment etc provide evidence of evidence-based medicine for Clinical application.

DETAILED DESCRIPTION:
RPH is a new therapy for hemorrhoid following the improvement of rubber band ligation.RPH +Simplified Milligan-Morgan is one of important means of modern surgery.The operation method was improved and developed on the basis of Chinese medicine traditional loop ligature and it also embodies uniqueness and advantage of the treatment of mixed hemorrhoids combined traditional Chinese and Western Medicine.The study intends to compare five surgery ways through 3000 cases of patients with mixed hemorrhoid from 12 hospitals,observing the efficacy and safety of various operative methods.Exploration of RPH + Simplified Milligan-Morgan operation indication, contraindication, operation steps and key points, and the operation complications and sequelae and treatment etc provide evidence of evidence-based medicine for Clinical application.

Diagnosis of all mixed hemorrhoids included in this study were performed according to"TCM anorectal diseases treatment guidelines" (2012 Edition) issued and implemented by the China Association of traditional Chinese Medicine .In all cases, the sub center for the unit, stratified by gender, age and disease.In every layer all cases were divided into 5 groups with random number table.Take balance check when test cases reach 80% of a predetermined number .If unbalanced index is larger , the following cases should be assigned according to the principle of the imbalance index reduction.All the cases were assigned to five groups in accordance with experiment design methods of random, contrast ,balance, parallel, and multicenter.Each sub center, each test group has 50 patients.

All the cases involved conducted corresponding preoperative examination and evaluation, respectively using 5 kinds of predetermined operation after grouping.Patients are in strict accordance with the "gynecology of traditional Chinese medicine" (Second Edition) for perioperative treatment in the preoperative, intraoperative and postoperative .

Observation indexes of this study include:General observation index,effective observation index,Safety observation index and severe adverse events.All the data use Excel to establish the data set ,analyzed by SPSS21.0.

ELIGIBILITY:
Inclusion Criteria:

* Conform to the diagnosis standard of mixed hemorrhoid
* Internal hemorrhoids indexing for II, III and IV
* Male or female,at the age of 18 to 65 years old
* No previous history of rectum and anus surgery
* Consent to treatment scheme in this study and sign informed consent

Exclusion Criteria:

* Under the age of 18 and Age more than 65 years.
* Combine with other colorectal anal diseases:tumor、crohn's disease、Ulcerative colitis, intestinal tuberculosis, anal fissure, anal fistula and perianal abscess etc.
* Combine with severe heart and brain blood vessels, liver, kidney and blood system diseases.
* Allergic or scar constitution.
* Pregnancy and lactation period or during menstruation.
* Mental illness or mental retardation, unclear expression .
* Other factors that may affect the results of the study or testers who should not enter the test according to researchers' judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
operative time | 1 day
  Effective observation index will be assessed by the operative time.
postoperative hospital stay | participants will be followed for the duration of hospital stay, an expected average of 1 weeks
  Effective observation index will be assessed by the postoperative hospital stay.
bloody stool | up to 6 months
  Effective observation index will be assessed by the bloody stool.
anal pain | up to 6 months
  Effective observation index will be assessed by the bloody stool.
sensation of rectal tenesmus | up to 6 months
  Effective observation index will be assessed by the sensation of rectal tenesmus.
Internal hemorrhoids prolapse | up to 6 months
  Effective observation index will be assessed by the Internal hemorrhoids prolapse.
External hemorrhoids swelling | up to 6 months
  Effective observation index will be assessed by the External hemorrhoids swelling.
Epicanthus situation | up to 6 months
  Effective observation index will be assessed by the Epicanthus situation.
postoperation hemorrhage | up to 6 months
  Safety observation index will be assessed by the postoperation hemorrhage.
postoperative uroschesis | up to 6 months
  Safety observation index will be assessed by the postoperative uroschesis.
rectovaginal fistula | up to 6 months
  Safety observation index will be assessed by the rectovaginal fistula.
Secondary anal fissure | up to 6 months
  Safety observation index will be assessed by the Secondary anal fissure.
postoperative perianal haematoma or thrombosis | up to 6 months
  Safety observation index will be assessed by the postoperative perianal haematoma or thrombosis.
fecal incontinence | up to 6 months
  Safety observation index will be assessed by the fecal incontinence.
anorectal stenosis | up to 6 months
  Safety observation index will be assessed by the anorectal stenosis.

SECONDARY OUTCOMES:
General observation index(composite) | 2 days
  General condition:sex.age.height.weight etc.and heart rate, pulse,respiration ,blood pressure etc.

OTHER OUTCOMES:
Severe adverse events | up to six months

CONTACTS AND LOCATIONS:
Overall Officials: Hu Fan, postgraduate, Principal Investigator — mentoring relationship; Hu Hua, postgraduate, Principal Investigator — Mentoring relationship
Locations (12):
- China (12):
  - The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine, Hefei, Anhui
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - Eighth Hospital of Wuhan City, Wuhan, Hubei
  - Changde Hospital of Hunan University of Traditional Chinese Medicine, Changde, Hunan
  - Changsha Hospital of Hunan University of Traditional Chinese Medicine, Changsha, Hunan
  - The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine, Changsha, Hunan
  - The Second Affiliated Hospital of Hunan University of Traditional Chinese Medicine, Changsha, Hunan
  - Chenzhou Hospital of Southern Medical University, Chenzhou, Hunan
  - Yueyang Hospital of Hunan University of Traditional Chinese Medicine, Yueyang, Hunan
  - The Third Affiliated Hospital of Nanjing University of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Xuzhou Hospital of Nanjing University of Traditional Chinese Medicine, Xuzhou, Jiangsu
  - Teaching Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan